CLINICAL TRIAL: NCT03603249
Title: Trimetazidine as an Adjunct to Enhance Clopidogrel Response: The TRACER Study.
Brief Title: Trimetazidine as an Adjunct to Enhance Clopidogrel Response.
Acronym: TRACER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CEC170/04/16
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-07

CONDITIONS: Platelet Dysfunction Due to Drugs
Keywords: platelet inhibition; platelet reactivity; clopidogrel; trimetazidine
MeSH Terms: interventions — Trimetazidine

STUDY DESIGN:
Intervention Model Description: The study will be of a prospective, randomized, controlled, sequential trial design.
Masking Description: The Outcomes Assessor will be independent of the Clinical Research Associates, i.e. he/she will be analyzing the VerifyNow samples without knowledge of the intervention the patient has received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clopidogrel and Trimetazidine Arm (Experimental): Patients on DAPT for at least 6 months will be tested for platelet function testing with the P2Y12 VerifyNow assay at baseline. The patients will then undergo at least a 2-week course of Trimetazidine 35 mg/q12h, followed thereafter by platelet function testing.
  Interventions: Drug: Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine — Trimetazidine is a clinically effective antianginal agent that has no negative inotropic or vasodilator properties (6). It is presently clinically used throughout Europe and in >80 countries worldwide. It is a cytoprotective drug that normalizes metabolic disturbances in low-flow ischemia via several-not yet fully understood-mechanisms of action (7). The best-known mechanism of action is its capacity to inhibit β-oxidation of free fatty acid (FFA) (7).
  Other Names: Vasteral MR, Laboratoires Servier, France

SUMMARY:
Hypothesis:

Trimetazidine improves Clopidogrel response in patients.

• The investigators postulate that the inhibition of platelet aggregation in response to Clopidogrel may be accentuated by Trimetazidine, i.e. Trimetazidine enhances Clopidogrel response.

Null Hypothesis:

There is no difference in Clopidogrel response in patients with stable coronary artery disease with adjunctive Trimetazidine.

DETAILED DESCRIPTION:
Rationale and Background:

Dual antiplatelet therapy with Aspirin and Clopidogrel represents the standard of care for the prevention of recurrent ischemic events in patients undergoing percutaneous coronary intervention (PCI). For more than 10 years, dual antiplatelet therapy with Aspirin and Clopidogrel has remained the cornerstone of treatment for patients with acute coronary syndrome (ACS). However, some patients have impaired Clopidogrel response and thus persist with high on-treatment platelet reactivity (HOT-PR) resulting in an increased risk of atherothrombotic events (1). This can be attributed to several factors such as genetic polymorphisms regulating the activity of the cytochrome P450 (CYP) 2C19 enzyme, which is key in metabolizing Clopidogrel into its active metabolite (2,3). The boxed warning added to the Clopidogrel label underscoring the potential risk of adverse cardiovascular outcomes among patients with a "poor metabolizer" genotype and advocating the use of other antiplatelet medications or alternative dosing strategies for these patients (4) has led to investigations of treatment options associated with more optimal platelet inhibition. These include increasing Clopidogrel dosing, adding a third antiplatelet agent (e.g. Cilostazol) and switching to a novel generation P2Y12 inhibitor (e.g. Prasugrel or Ticagrelor). The novel oral P2Y purinoceptor 12 (P2Y12) receptor inhibitors Prasugrel and Ticagrelor were approved by the FDA for clinical use in 2009 and 2011 respectively (5).

Activation of P2Y12 inhibits AC, causing a decrease in cAMP and VASP-P levels and activation of P2Y1 causes an increase in intracellular Ca2+ levels. These changes promote platelet aggregation by altering the ligand-binding properties of the GP IIb/IIIa receptor. Inhibition of the P2Y12 receptor therefore, suppresses platelet activation (5).

Trimetazidine is a clinically effective antianginal agent that has no negative inotropic or vasodilator properties (6). It is presently clinically used throughout Europe and in >80 countries worldwide. It is a cytoprotective drug that normalizes metabolic disturbances in low-flow ischemia via several-not yet fully understood-mechanisms of action (7). The best-known mechanism of action is its capacity to inhibit β-oxidation of free fatty acid (FFA) (7). The main cytoprotective mechanisms (7) are outlined in the following table:

FFA breakdown inhibition and glucose breakdown stimulation Reduction in the amount of oxygen necessary for ATP production Reduction in the cellular accumulation of lactic acid and H+ Reduction in the cellular accumulation of Na+ and Ca2+ Reduction in ATP losses for maintaining ion homeostasis Reduction of adverse effects of overloading cells with calcium Anti-radical effect Reduction of granulocyte infiltration to the ischaemic and reperfused area of the myocardium Cardiomyocyte apoptosis inhibition

Trimetazidine prevents a decrease in intracellular ATP levels, thereby ensuring the proper functioning of ionic pumps and transmembrane sodium-potassium flow whilst maintaining cellular homeostasis (8). It is also known that ATP acts as an antagonist of the effects of ADP at P2Y1 and P2Y12 receptors (9,10) and that high concentrations can inhibit ADP-induced platelet aggregation (11,12). The drug is suitable for initial use as monotherapy in patients with angina pectoris and because of its different mechanism of action as adjunctive therapy in those with symptoms not sufficiently controlled by nitrates, beta blockers or calcium channel antagonists. Multicenter trials of Trimetazidine by a European collaborative working group have demonstrated that the antianginal efficacy of Trimetazidine is equivalent to that of propranolol but does not reduce cardiac rate-pressure product or coronary blood flow (13). The 2013 European Society of Cardiology (ESC) guidelines take into consideration the possibility of using Trimetazidine as treatment for stable coronary artery disease-however, this is a IIb recommendation (14). The current recommendations do not consider this treatment in other cardiovascular diseases such as chronic heart failure (15) or acute coronary syndromes (16,17). The role of Trimetazidine in other coronary conditions has yet to be clearly established (18).

Trimetazidine has been treated as a drug with a high safety and tolerability profile (19). It has been generally very well tolerated in clinical trials and usually only isolated cases of adverse events (ADRs-adverse drug reactions) were observed during treatment (mainly gastrointestinal disturbances e.g. vomiting, nausea) (7). Some other very rare and reversible adverse effects have also been described such as thrombocytopenia, agranulocytosis and liver dysfunction (20). Other minor adverse effects e.g. headache were also reported. Most of them were not considered to be directly related to Trimetazidine (20). However, some recently reported ADRs require careful evaluation in longer follow-up. The main identified serious ADR is connected to Parkinson's syndrome and related symptoms such as tremor (21). It is worth emphasizing that extrapyramidal symptoms reported in patients receiving Trimetazidine have a very low prevalence (incidence of 0.36/100,000 person-years) and are generally reversible after drug withdrawal.

The investigators postulate that the inhibition of platelet aggregation in response to Clopidogrel may be accentuated by Trimetazidine, i.e. Trimetazidine enhances Clopidogrel response.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 and 74 years of age,
2. have stable coronary artery disease, already on DAPT with aspirin and clopidogrel for at least 6 months,
3. not on any physician-prescribed medications or complementary/alternative therapies,

Exclusion Criteria:

1. presence of active internal bleeding or history of bleeding diathesis or clinical findings associated with an increased risk of bleeding,
2. history of ischemic or hemorrhagic stroke, transient ischemic attack, intracranial neoplasm, arteriovenous malformation, or aneurysm,
3. clinical and/or hemodynamic instability,
4. within 1 month of placement of a bare metal stent,
5. within 30 days of coronary artery bypass graft surgery or PCI without a stent placed,
6. planned coronary revascularization,
7. treatment with fibrin-specific fibrinolytic therapy <24 h or non-fibrin-specific fibrinolytic therapy <48 h,
8. use of an oral anticoagulation agent or international normalized ratio >1.5,
9. body weight <60 kg,
10. age >75 years,
11. hemoglobin <10 g/dL,
12. platelet count <100×106/μL,
13. creatinine >2 mg/dL,
14. hepatic enzymes >2.5 times the upper limit of normal,
15. pregnancy and/or lactation.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Platelet Reactivity Units at baseline compared to post-intervention with Trimetazidine | 10-14 days
  The investigators postulate that inhibition of platelet aggregation in response to Clopidogrel may be accentuated by Trimetazidine, i.e. Trimetazidine enhances Clopidogrel response.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of the West Indies, Saint Augustine, North, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: Yes
All available data can be obtained by contacting the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Throughout the entire study duration.
Access Criteria: Unrestricted

REFERENCES:
- [Derived] Seecheran N, Seebalack V, Seecheran R, Maharaj A, Boodhai B, Seecheran V, Persad S, Motilal S, Tello-Montoliu A, Schneider D. TRimetazidine as an Agent to affeCt clopidogrEl Response: The TRACER Study. Cardiol Ther. 2019;8(2):229-237. doi: 10.1007/s40119-019-0139-0. Epub 2019 Jul 10. PMID 31292901